CLINICAL TRIAL: NCT05381233
Title: Quality of Life and Functional Performance in Children With Spastic Cerebral Palsy in Relation to Care Burden and Fatigue of Their Mothers
Brief Title: Quality of Life and Functional Performance in Children With Spastic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sara Shawki Mohamed (Other)
Responsible Party: Sponsor-Investigator, Sara Shawki Mohamed, assistant lecturer, October 6 University
Organization: October 6 University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 78093
Record Dates: First submitted 2022-04-04; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Evaluations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hemiplegic group (Other): hemiplegic patient
  Interventions: Other: Gross motor function classification System (GMFCS); Other: Arabic Version of Zarit burden Inventory measure; Other: Arabic Version of Chalder Fatigue Scale (CFQ version 11)
- Group diaplegic (Other): diaplegic patient
  Interventions: Other: Gross motor function classification System (GMFCS); Other: Arabic Version of Zarit burden Inventory measure; Other: Arabic Version of Chalder Fatigue Scale (CFQ version 11)
- group quadriplegic (Other): quadriplegic patient
  Interventions: Other: Gross motor function classification System (GMFCS); Other: Arabic Version of Zarit burden Inventory measure; Other: Arabic Version of Chalder Fatigue Scale (CFQ version 11)

INTERVENTIONS:
Other: Gross motor function classification System (GMFCS) — assessment
Other: Arabic Version of Zarit burden Inventory measure — assessment
Other: Arabic Version of Chalder Fatigue Scale (CFQ version 11) — assessment

SUMMARY:
Caregiver Burden (CB) is expressed as a multidimensional response related to caregiving, including physical, psychological, emotional, social, and economic problems and has been identified as a public health concern. All these factors negatively affect caregiver health and indirectly affect the care of the disabled child .To provide better support for parents of children with CP, we must understand the difficulties faced those parents and identify the key and common areas where assistance can be rendered.

DETAILED DESCRIPTION:
The symptoms of CP vary from person to person. A person with severe CP might need to use special equipment to be able to walk, or might not be able to walk at all and might need lifelong care. A person with mild CP, on the other hand, might walk a little awkwardly, but might not need any special help. CP does not get worse over time, though the exact symptoms can change over a person's lifetime.

ELIGIBILITY:
Inclusion Criteria:

* Age older then 18 years.
* there BMI will be ranged from 18.5 too 24.9 kg/m2 (Misra et al., 2009) .
* They are the main caregiver for there children.
* They are of low or middle socioeconomic status according too socioeconomic status scale (El-Gilany et al., 2012).
* Having at least 7months of experience in taking care of the child.
* They have no congenital spinal anomalies or lower limb deformities.

Exclusion Criteria:

* Children wif congenital anomalies and chromosomal disease.
* Children wif recent musculoskeletal surgery.
* Any associated problems.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Gross motor function classification System (GMFCS) | 3 months
  Which are a Standardized method too, classify gross motor function in children with (CP) aged from 2 too, 18years. Teh GMFCS are a 5-level system designed too, reflect differences in gross motor function that are meaningful in teh daily lives of children with CP and there families, with an emphasis on sitting and walking. A classification are made by determining which level best corresponds too, a child"s present gross motor function (Palisano et al., 1997). dis scale will be used for detecting teh CP child functional performance level
Arabic Version of Zarit burden Inventory measure | 3 months
  It are one of the most commonly used measures of caregiver burden (Knight et al., 2000). The care burden of all the participants will be evaluated by the Zarit burden Inventory measures (ZBI). The ZBI assesses the stress suffered by those whom give care too the persons in need. Initially developed and validated more TEMPthan 25 years ago (Zarit et al., 1980)

CONTACTS AND LOCATIONS:
Overall Officials: emad ismaiel, phd, Study Director — physical therapy
Locations (1):
- Emad, Cairo, Egypt